CLINICAL TRIAL: NCT00170833
Title: A Prospective, Multicenter, Open Label, Randomized Study of the Safety, Tolerability and Efficacy of Everolimus (RAD001) With Basiliximab, Corticosteroids and Lower Levels Versus Higher Levels of Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: Safety, Tolerability and Efficacy of Everolimus With Lower Versus Higher Levels of Tacrolimus in de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AUS09
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Renal/Kidney, transplantation, everolimus, calcineurin sparing
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
This study will assess the safety and efficacy of everolimus with basiliximab, corticosteroids and lower levels versus higher levels of tacrolimus in de novo renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 65 years of age
* Male or female patients who are primary cadaveric, living unrelated or non-HLA identical living related donor renal transplant recipients
* The renal cold ischemic time (CIT) must be < 30 hours
* The age of the donor must be between 10 and 59 years and not meet UNOS expanded donor criteria

Exclusion criteria

* Patients meeting any of the following criteria at baseline will be excluded from study participation.
* Patients who have previously received an organ transplant
* Patients who are recipients of a multiple organ transplants
* Recipients of non heart-beating donor organs

Other protocol define inclusion/exclusion criteria may apply. Patients who are recipients of A-B-O incompatible transplants or T-cell crossmatch positive transplants Patients with current panel reactive T-cell antibodies (PRA) titers of 50% or more (when the test is performed with dithiothreitol treated patient's serum) Patients who are known to have a positive hepatitis C serology, who are human immunodeficiency virus (HIV) or Hepatitis B surface antigen positive. Laboratory results obtained within 6 months prior to first dose of everolimus are acceptable. Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C are excluded Presence of cardiac disease ( Old New York Heart Association Classification Grade 3, elevated creatine phosphokinase myocardial binding isoenzyme (CPK-MB)or any cardiac disease considered to be unsafe for the study by the investigator) 10.Presence of severe hypercholesterolemia ( 350 mg/dL, 9.1 mmoL/dL) or hypertriglyceridemia ( 500mg/dL, 5.6 mmoL/L). Patients with controlled hyperlipidemia are acceptable 11.White blood cell (WBC) count 4500/mm3, or platelet count 100,000/mm3 12.Evidence of liver injury as indicated by an abnormal liver profile (AST, ALT, alkaline phosphatase or total bilirubin 3 times ULN) before transplantation 13.Presence of any severe allergy requiring acute (within 4 weeks of baseline) or chronic treatment, or hypersensitivity to drugs similar to everolimus (e.g., macrolides) 14.The use of any investigational drug within 4 weeks of the baseline period 15.Patients who have been treated with non-protocol immunosuppressive drug or treatment within 1 month prior to first dose of everolimus 16.Patients with severe systemic infections 17.Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator, preclude enrollment in this trial 18.Malignancy (current or history within last 5 years) except for successfully treated localized basal or squamous cell carcinoma of the skin 19.Patients with any medical condition requiring long-term anticoagulation, such as heparin, low molecular weight heparin, or warfarin, after transplantation (Low dose aspirin, clopidogrel, or cilostazol treatment is allowed) 20.Abnormal physical or laboratory findings of clinical significance within 2 weeks prior to first dose of everolimus which at investigators discretion would interfere with the objectives of the study 21.Breast feeding women 22.Patients with symptoms of significant somatic or mental illness. Unresolved history of drug or alcohol abuse 23.Inability to cooperate or communicate with the investigator 24.Donors that meet the UNOS expanded donor criteria

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-11; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
renal function as measured by serum creatinine at 6 months post-transplant

SECONDARY OUTCOMES:
Renal function as measured by calculated creatinine clearance and calculated glomerular filtration rate at 6 months
Occurrence of biopsy-proven acute rejection at 6 months post-transplant
Combined and individual incidence of biopsy-proven acute rejection episodes, graft loss, and death at 6 months
Incidence of adverse events and serious adverse events
Incidence of New Onset Diabetes post-transplant at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Derived] Chan L, Greenstein S, Hardy MA, Hartmann E, Bunnapradist S, Cibrik D, Shaw LM, Munir L, Ulbricht B, Cooper M; CRADUS09 Study Group. Multicenter, randomized study of the use of everolimus with tacrolimus after renal transplantation demonstrates its effectiveness. Transplantation. 2008 Mar 27;85(6):821-6. doi: 10.1097/TP.0b013e318166927b. PMID 18360262